CLINICAL TRIAL: NCT00865319
Title: A Multicenter Phase 2 Study Comparing 99m Tc EC-DG SPECT/CT With 18F FDG PET/CT in the Evaluation of Patients With Non-small Cell Lung Cancer (NSCLC)
Brief Title: Phase 2 Study Comparing 99mTc-EC-DG SPECT/CT With 18F FDG PET/CT in Patients With Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cell>Point LLC (Industry)
Collaborators: Numoda (Industry); Venn Life Sciences (Other); Camargo Pharmaceutical Services (Industry); Biomedical Services (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-05-232 Amendment 1
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Spect CT Imaging; PET CT Imaging as Comparator
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 99 m Tc-EC-DG (Experimental): 99m Tc-Ec-DG injection followed by SPECT/CT imaging (range 20-30 mCi) 1mg EC-DG
  Interventions: Radiation: Radiolabeled (99Tc) EC-DG (ethylenedicysteine-deoxyglucose)
- 18F-FDG (Active Comparator): 18 F FDG injection followed by PET/CT imaging
  Interventions: Radiation: 18 F fluorodeoxyglucose

INTERVENTIONS:
Radiation: Radiolabeled (99Tc) EC-DG (ethylenedicysteine-deoxyglucose) — one injection of Technetium ethylenedicysteine-deoxyglucose to yield a target activity of 20mCi (range 20-30 mCi) to be given by slow IV push (over 3-5 minutes) 1mg of EC-DG to be injected
  Arms: 99 m Tc-EC-DG
Radiation: 18 F fluorodeoxyglucose — single injection of 18F FDG (range 10-20mCi)
  Arms: 18F-FDG

SUMMARY:
This is a multiple-center Phase 2 study designed to expand the patient safety and clinical information using 99m Tc-Ec-DG with Spect/CT imaging, to develop procedures and methods for evaluation of the imaging studies, to determine comparability of diagnostic information between SPECT and SPECT/CT imaging and to to compare the safety and efficacy of 99m Tc-EC-DG SPECT/CT with 18F-FDG PET/CT in imaging patients with biopsy confirmed diagnosis of Non-small Cell Lung Cancer.

DETAILED DESCRIPTION:
Male and female patients at least 18 years of age with untreated Non-small Cell Lung Cancer who have non-incisional biopsy definitive evidence of disease (or from cytology results from a bronchoscope procedure) and who have been previously certified (per centers for Medicare and Medicaid Services requirements) by their physicians will be consented for the study. The study consists of a screening visit, gold-standard 18F-FDG PET/CT imaging followed by the investigational agent 99m Tc-Ec-DG SPECT/CT. The study procedures can be performed within 5-7 days of signing the informed consent. [To better meet the standard of care at each clinical location, the PET/CT can be performed as part of pre-study procedures on a PET/CT camera previously qualified by the site to meet the standards required for the study. If this occurs, the SPECT/CT must be performed within 45 days of the PET/CT imaging procedures.] Patients will be seen 24 hours after the 99m Tc-Ec-DG injection for safety. A 21-day follow-up period (after the SPECT/CT image) will allow the investigator to acquire additional imaging, surgical, pathology and treatment documentation. [An actual patient visit is NOT required at the 21-day follow-up time point.]

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years old;
* Have non-incisional biopsy demonstrating definitive evidence for NSCLC (Cytology results confirming NSCLC from a bronchoscope procedure will also be acceptable) and have not been treated for lung cancer (surgery, radiation and/or chemotherapy); A copy of the actual report must be requested by the patient through a medical release form if not already done. The copy must be available to the study doctor within 28 days of the screening visit/ Visit 1 ;
* Be certified as per centers for Medicare and Medicaid Services (CMS) requirements and be eligible for a PET scan;
* Have an Eastern Co-operative Oncology Group (ECOG) performance rating ≤ 2 (see Appendix 1);
* Males or non-pregnant, non-lactating females who are postmenopausal, naturally or surgically sterile, or who agree to use effective contraceptive methods throughout the course of the study. Postmenopausal is defined as at least 12 months natural spontaneous amenorrhea, or at least 6 weeks following surgical menopause (bilateral oophorectomy);
* Females of childbearing potential and males with female sexual partners of childbearing potential must agree to use one of the following acceptable birth control methods:

  1. Surgically sterile (hysterectomy or bilateral oophorectomy);
  2. Surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to study initiation). Documentation is required;
  3. Intrauterine device (IUD) in place for at least 3 months;
  4. Double-barrier method (condom and diaphragm) with spermicide for at least 14 days prior to screening and through study completion;
  5. Stable hormonal contraceptive (oral, topical, vaginal or implanted/injected) for at least 3 months prior to study and through study completion;
  6. Abstinence;
  7. Single-barrier method for at least 14 days prior to screening and though study completion for vasectomized males or females with vasectomized partners;
* Have a fasting blood glucose of less than 200 mg/dL at screening;
* Have reported clinical symptoms consistent with a confirmed diagnosis of NSCLC;
* BE able to tolerate SPECT/CT and PET/CT imaging. This includes:

  * Laying in the same position without moving for approximately 45 minutes;
  * Able to tolerate a claustrophobic area;
  * Ability to hold their arms overhead for approximately 45 minutes;
* Be able to fast prior to SPECT/CT and PET/CT imaging, with length of fasting dependent on the time of the scan (or follow site specific fasting and/or diet restrictions):

  * A morning scan (08:00-12:00) will require fasting from midnight;
  * An afternoon scan (12:00-onward) will require a minimum 6 hour fast;
* Be able to eat a high protein/low carbohydrate meal as the last meal before SPECT/CT and PET/CT imaging (or follow site specific fasting and/or diet restrictions);
* Be able to make the scheduled appointments within the designated time windows (PET/CT imaging within 7 days of qualifying for the study, the second imaging session with SPECT/CT imaging 1 - 3 days after the initial imaging visit, with at least 24 hours between PET/CT and SPECT/CT imaging). If the PET/CT was done as part of the pre-screening procedures and was conducted on a previously qualified PET camera for the study, the SPECT/CT must be done within 45 days of the PET/CT imaging procedures;
* Have safety laboratory values that in the opinion of the Investigator do not place the patient at undue risk if the patient were to participate in the study. This includes (but is not limited to):

  * Alanine aminotransferase 2.5 × upper limit of normal (ULN);
  * Aspartate aminotransferase 2.5 × ULN;
  * Creatinine 2.5 × ULN;
  * Bilirubin 2.0 × ULN;
* Able to understand and provide signed informed consent;
* Females of childbearing potential must have a negative urine or serum β-human chorionic gonadotropin (hCG) pregnancy test at screening.

Exclusion Criteria:

* Any clinically significant safety concerns (laboratory, electrocardiogram [EKG], physical examination, other) that, in the opinion of the Investigator, would place the patient at undue risk if the patient were to participate in the study;
* Undergoing any current treatment for cancer (radiation therapy, surgery or chemotherapy);
* Diabetic with insulin dependence (Patients who have a known insulin dependence for diabetes can be included in the study if the standard of care protocol in place at the clinical site provides for the management of the patient's glucose level sufficiently to allow the PET/CT imaging to be performed. The same glucose management used for the PET/CT imaging should be applied to the SPECT/CT imaging procedures. A waiver will be required to be completed by the clinical site and approved by the sponsor or designee;
* Patient weight above the SPECT/CT and PET/CT table weight limit;
* Failure to have a non-incisional biopsy definitive diagnosis for NSCLC (or cytology report from a bronchoscope); [a copy of the biopsy/cytology report must be available to the investigator within 28 days of Visit 1];
* Will not agree to use an effective means of contraception for the duration of the study (males and females);
* Known hypersensitivity to EC-DG or FDG or similar compounds including any of the inactive ingredients;
* Known or suspected pregnancy, lactation or planned pregnancy (females and male partners);
* Clinically significant mental illness (to be determined by the Investigator);
* Exposure to any investigational agent within 30 days prior to screening visit or participating in an ongoing clinical study (this criteria can be overruled by the Principal Investigator with appropriate documentation of the reason for the exception);
* Patient has a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety: Through adverse event collection | from 99m Tc-Ec-DG injection through 21 days

SECONDARY OUTCOMES:
Efficacy: Comparison of 18F FDG PET/CT image against 99m Tc-EC-DG image | End of study
Efficacy: determine comparability of diagnostic information between SPECT (acs) and SPECT/CT (als) imaging | End of Study
Efficacy: To provide evidence of 99m Tc-Ec-DG in identifying anatomical regions with known Non-small cell lung cancer and in determining extent of disease in these patients as compared to 18F-FDG PET/CT imaging | End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Donald Blaufox, MD, Principal Investigator — Albert Einstein University, Montefiore Medical Center
Locations (6):
- United States (5):
  - Baptist Health South Florida, Coral Gables, Florida
  - Decatur Memorial Hospital Department of Radiology, Decatur, Illinois
  - John Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Division of Nuclear Medicine, Rochester, Minnesota
  - Montefiore Medical Center, Department of Nuclear Medicine, The Bronx, New York
- Lions Gate Hospital, North Vancouver, British Columbia, Canada

REFERENCES:
- See also: Location of the study — http://mayoclinic.com
- See also: Sponsor Link — http://cellpointweb.com
- See also: Clinical Site — http://www.montefiore.org
- See also: Clinical Site — http://www.baptisthealth.net
- See also: Clinical Site — http://www.dmhcares.org